CLINICAL TRIAL: NCT07211178
Title: Evaluating Minimal Residual Disease (MRD) Through Longitudinal Circulating Tumor DNA (ctDNA) Profiling in Breast Malignancies
Acronym: GEMINI Breast
Status: Recruiting | Type: Observational
Sponsor: Tempus AI (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-CA-010
Record Dates: First submitted 2025-09-19; First posted 2025-10-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; TNBC - Triple-Negative Breast Cancer; HR Positive/HER-2 Negative Breast Cancer; HER2 + Breast Cancer; Early Stage Breast Cancer
Keywords: Minimal Residual Disease; MRD; Next generation sequencing; NGS; ctDNA; Early Stage Breast Cancer; TNBC - Triple Negative Breast Cancer; HR positive / HER-2 negative breast cancer; HER2+ breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva, blood and leftover tissue will be collected in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Neoadjuvant Therapy: There are no interventions in this observational study. Cohort 1 includes participants who will receive neoadjuvant treatment prior to surgery.
  Interventions: Other: There are no interventions in this observational study.
- Cohort 2: Adjuvant Therapy / Surveillance: There are no interventions in this observational study. Cohort 2 includes participants who will receive adjuvant therapy after surgery.
  Interventions: Other: There are no interventions in this observational study.
- Cohort 3: 5 Years Post-Diagnosis Surveillance: There are no interventions in this observational study. Cohort 3 includes participants who have no evidence of disease for at least 5 years post diagnosis.
  Interventions: Other: There are no interventions in this observational study.

INTERVENTIONS:
Other: There are no interventions in this observational study. — There are no interventions in this observational study.

SUMMARY:
For patients with breast cancer, it's important to find any remaining cancer cells after they've had their main treatment. Even a few cells, called minimal residual disease (MRD), can lead to the cancer coming back later.

A way to find these cells is by looking for tiny bits of cancer DNA that are shed into the blood. This is called circulating tumor DNA (ctDNA). A simple blood test, often called a liquid biopsy, can detect this ctDNA. This research aims to see if finding this cancer DNA in the blood can help predict if a patient's cancer will return. It also may help find out if the treatment is working.

Ultimately, the results of this research may help doctors better manage breast cancer and develop new and improved tests and treatments.

ELIGIBILITY:
Inclusion Criteria:

All Cohorts:

1. Willing and able to participate in the research and provide biospecimens
2. Willing and able to provide informed consent
3. Must be diagnosed with breast cancer

Cohort 1: Neoadjuvant Treatment Cohort 1A: Newly Diagnosed, High Risk HR+,HER2-

1. A known or suspected HR+, HER2- breast cancer treated with curative intent (Stage II to III disease)
2. Patients are considered at high risk of recurrence, defined as 4 or more positive axillary lymph nodes (ALNs), or between 1-3 positive ALNs and either grade 3 disease or tumor size of 5 cm or larger.

Cohort 1B: HER2+ 1. A known or suspected HER2+ breast cancer treated with curative intent (Stage II to III disease). Inclusive of HR+ or HR- patients.

Cohort 1C: Triple Negative Breast Cancer

1. A known or suspected triple negative breast cancer treated with curative intent (Stage I to III disease).

Cohort 2: Adjuvant Therapy / Surveillance Cohort 2A: Newly Diagnosed HR+,HER2-

1. A known or suspected HR+, HER2- breast cancer treated with curative intent (Stage II to III disease)
2. Patients are considered at high risk of recurrence, defined as 4 or more positive axillary lymph nodes (ALNs), or between 1-3 positive ALNs and either grade 3 disease or tumor size of 5 cm or larger.
3. Have undergone curative intent surgery with no clinical evidence of disease.

Cohort 2B: HER2+

1. A known or suspected HER2+ breast cancer treated with curative intent (Stage II to III disease)
2. Have undergone curative intent surgery with no clinical evidence of disease.

Cohort 2C: Triple Negative Breast Cancer

1. A known or suspected triple negative breast cancer treated with curative intent (Stage I to III disease)
2. Have undergone curative intent surgery with no clinical evidence of disease.

Cohort 3: 5-Years Post-Diagnosis Surveillance (NED)

1. A known HR+, HER2- breast cancer treated with curative intent (Stage II to III disease).
2. No Evidence of Disease (NED) ≥ 5 years from initial diagnosis.
3. Patients are considered at high risk of recurrence, defined as 4 or more positive axillary lymph nodes (ALNs), or between 1-3 positive ALNs and either grade 3 disease or tumor size of 5 cm or larger.

Exclusion Criteria:

1. Not willing or able to adhere with the study procedures
2. Active secondary malignancy
3. Diagnosis of a malignancy within 3 years of breast cancer diagnosis Note: Ductal carcinoma in situ (DCIS, ipsilateral or contralateral) within 3 years is not excluded.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of this study includes early stage breast cancer patients with triple negative breast cancer (Stages I to III), HER2 positive (Stages II and III), and high risk HR positive HER-2 negative (Stages II and III).
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease-Free Survival (iDFS) stratified by MRD status during neoadjuvant, post-surgery landmark, post definitive treatment (surveillance), and long-term follow-up | 5 years

SECONDARY OUTCOMES:
Distant disease free survival rates stratified by MRD status during neoadjuvant treatment | 5 years
Overall Survival rates stratified by MRD status during neoadjuvant treatment, post-surgery landmark, post definitive treatment (surveillance), and long-term follow-up | 5 years
Pathologic Complete Response (pCR) or Residual Cancer Burden (RCB) rate stratified by MRD status at post-surgery landmark | 5 years
Time from First Positive MRD Sample to Recurrence | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Ting-Lin, MD, Principal Investigator — Tempus AI
Locations (1):
- PIH Health Whittier Hospital, Whittier, California, United States